CLINICAL TRIAL: NCT01457729
Title: Telemedizinisches Trainings-Monitoring Von Patienten Mit Obstruktivem Schlafapnoesyndrom
Brief Title: Ergometer Training in Patients With OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Pneumologie Hagen Ambrock eV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERGO2011
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: ergometer; training; motivation; telemonitoring; sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Motivation (No Intervention): Patients are asked to complete a telemonitored Ergometer training for 4 Weeks, at least 30 minutes per day, no more intervention is done.
- Motivation (Other): Patients are asked to complete a telemonitored Ergometer training for 4 Weeks, at least 30 minutes every day. If training time declines to less than 20 minutes per day for one week, a motivation phone call will take place once a week.
  Interventions: Behavioral: Motivation by Telephone Call

INTERVENTIONS:
Behavioral: Motivation by Telephone Call — Telephone call not exceeding 10 minutes according to a protocol
  Arms: Motivation

SUMMARY:
Patients with suspected OSA (obstructive sleep apnoea syndrome) are asked to use a standard bike ergometer which is additionally equipped with a system to gather training data and the ability to send daily training time to an internet server to which the physician has access. Training time of two groups is compared. Group one is not motivated while group two benefits from telephone feedback when training time declines. It is presumed that training time increases with better information and response to training behaviour.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected OSA
2. Capable of giving consent

Exclusion Criteria:

1. Symptomatic cardial infarction
2. Decompensated cardiac insufficiency
3. Hemodynamically effective cardiac arrhythmias
4. Hemodynamically significant Vitia (heart disease)
5. Insufficiently regulated arterial hypertension
6. Global respiratory insufficiency
7. Significant partial insufficiency (PAO2 <50mmHg or SaO2 < 80% at rest)
8. State after decompensation of Cor Pulmonale
9. Right ventricular strain at pulmonary hypertension at rest (pulmonary arterial pressure > 20 mmHg)
10. Severe osteoporosis
11. Higher degree of lung functional restriction: FEV1 <50% oder >60% of nominal value after bronchospasmolysis
12. Working performance on ergometer < 50%
13. Unstable bronchial asthma
14. Exacerbated COPD
15. Heavily overweight (BMI >40 or weight >140kg)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Training time | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karl Heinz Ruehle, Prof, Principal Investigator — Institut für Pneumologie Hagen Ambrock eV
Locations (1):
- Helios Klinik Hagen Ambrock, Hagen, North Rhine-Westphalia, Germany